CLINICAL TRIAL: NCT05291091
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of EDG-5506 on Safety, Biomarkers, Pharmacokinetics, and Functional Measures in Adults and Adolescents With Becker Muscular Dystrophy
Brief Title: Phase 2 Study of EDG-5506 in Becker Muscular Dystrophy (GRAND CANYON)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); ImagingNMD (Unknown); SYSNAV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDG-5506-201
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Adult Cohort 1 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten 10 mg; Drug: Placebo
- Adult Cohort 2 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten 10 mg; Drug: Placebo
- Adult Cohort 6 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten 10 mg; Drug: Placebo
- Adolescent Cohort 4 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten 5 mg; Drug: Placebo
- Adolescent Cohort 5 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten 12.5 mg; Drug: Placebo

INTERVENTIONS:
Drug: Sevasemten 10 mg — Sevasemten is administered orally once per day
  Arms: Adult Cohort 1; Adult Cohort 2; Adult Cohort 6
Drug: Sevasemten 5 mg — Sevasemten is administered orally once per day
  Arms: Adolescent Cohort 4
Drug: Sevasemten 12.5 mg — Sevasemten is administered orally once per day
  Arms: Adolescent Cohort 5
Drug: Placebo — Placebo is administered orally once per day

SUMMARY:
A study of sevasemten (EDG-5506) in Becker muscular dystrophy (known as CANYON) and pivotal cohort (known as GRAND CANYON). The EDG-5506-201 CANYON study was expanded to include an additional 120 adult participants in a cohort called GRAND CANYON, that is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of sevasemten in adults with Becker.

CANYON and GRAND CANYON are fully enrolled.

DETAILED DESCRIPTION:
The EDG-5506-201 protocol was amended to include an additional cohort thus consists of two parts.

Part 1: CANYON is a double-blind, randomized, placebo-controlled design to investigate the effect of sevasemten on the safety, pharmacokinetics, biomarkers, and functional measures. Approximately 32 adults and 18 adolescents with Becker muscular dystrophy are planned to enroll in this study. This study will have up to a 4-week Screening period, a 12-month Treatment period, followed by a 4-week follow-up period.

Approximately 32 adult participants will randomize to Cohort 1 or Cohort 2 in a 1:1 ratio then each cohort will further randomize to sevasemten or placebo in a 3:1 ratio.

Approximately 9 adolescent participants will enroll in Cohort 4 and randomize in a 2:1 ratio to sevasemten or placebo. Cohort 5 will randomize an additional 9 participants in a 2:1 ratio to either sevasemten or placebo after Cohort 4.

CANYON is now fully enrolled.

Part 2: GRAND CANYON or Cohort 6 is a double-blind, randomized, placebo-controlled design to investigate the safety and efficacy of sevasemten in adults with Becker muscular dystrophy after 18 months of treatment. Approximately 120 adults with Becker muscular dystrophy are planned to enroll in this study. This study will have up to a 4-week Screening period, an 18-month Treatment period, followed by a 4-week follow-up period.

Approximately 120 adult participants will be randomized in Cohort 6 in a 2:1 ratio either to sevasemten or placebo.

ELIGIBILITY:
The CANYON Study including the adolescent cohorts are fully enrolled.

GRAND CANYON eligibility is listed below.

Key Inclusion Criteria:

1. Adults (aged 18 to 50 years, inclusive) with a documented dystrophin mutation and phenotype consistent with Becker muscular dystrophy, and history of being ambulatory beyond 16 years of age without steroids; history of being ambulatory beyond 18 years of age with steroids.
2. Able to complete the 100-meter timed test in < 200 seconds with or without use of mobility aid devices.
3. Able to perform the North Star Ambulatory Assessment scale and achieve a score of 5 to 32, inclusive.

Key Exclusion Criteria:

1. Medical history or clinically significant physical examination/laboratory result that, in the opinion of the investigator, would render the participant unsuitable for the study. This includes contraindications to magnetic resonance imaging such as non-compatible implanted medical devices or severe claustrophobia.
2. Cardiac echocardiogram ejection fraction < 40%
3. Forced vital capacity predicted <60% or using daytime ventilatory support
4. Receipt of oral corticosteroids for the treatment of BMD in the previous 6 months.
5. Receipt of an investigational drug within 30 days or 5 half-lives (whichever is longer) of the screening visit in the present study.

Ages: 12 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 244 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events in those treated with sevasemten or placebo | 12 months (CANYON Cohorts 1, 2, 4, 5), 18 months (GRAND CANYON Cohort 6)
  All participants
Severity of adverse events in those treated with sevasemten or placebo | 12 months (CANYON Cohorts 1, 2, 4, 5), 18 months (GRAND CANYON Cohort 6)
  All participants
Change from Baseline in serum Creatine Kinase | 12 Months (CANYON Cohorts 1, 2)
  Adult participants
Change from Baseline in the North Star Ambulatory Assessment scale | 18 months (GRAND CANYON Cohort 6)
  Adult participants

SECONDARY OUTCOMES:
Change from Baseline in the protein fast skeletal muscle Troponin I | 12 months (CANYON Cohorts 1, 2), 18 months (GRAND CANYON Cohort 6)
  Adult participants
Change from Baseline in the North Star Ambulatory Assessment scale | 12 Months (CANYON Cohorts 1, 2)
  Adult participants
Change from Baseline in the North Star Assessment for Limb-Girdle Type Muscular Dystrophies scale | 12 Months (CANYON Cohorts 1, 2), 18 Months (GRAND CANYON Cohort 6)
  Adult participants
Change from Baseline in the 10-meter walk/run test | 12 Months (CANYON Cohorts 1, 2), 18 Months (GRAND CANYON Cohort 6)
  Adult participants
Change from Baseline in 100-meter timed test | 12 Months (CANYON Cohorts 1, 2), 18 Months (GRAND CANYON Cohort 6)
  Adult participants
Change from Baseline in stride velocity (95th percentile) | 18 Months (GRAND CANYON Cohort 6)
  Adult participants
Pharmacokinetics as measured by steady state plasma concentration | 12 Months (CANYON Cohorts 1, 2, 4, 5), 18 months (GRAND CANYON Cohort 6)
  All participants
Change from Baseline in growth as assessed by height centile on World Health Organization growth charts | 12 months (CANYON Cohorts 4, 5)
  Adolescent participants
Month 18 change from Baseline in fat fraction of upper leg muscles as assessed by Magnetic Resonance Imaging | 18 months (GRAND CANYON Cohort 6)
  Adult participants

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donovan, MD, PhD, Study Chair — Edgewise Therapeutics, Inc.; Roxana D. Dreghici, Study Chair — Edgewise Therapeutics, Inc.
Locations (51):
- United States (26):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - UC Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Rare Disease Research, LLC NC, Hillsborough, North Carolina
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - National Neuromuscular Research Institute, Austin, Texas
  - Neurology Rare Disease Center, Denton, Texas
  - Virginia Commonwealth University Health, Richmond, Virginia
- St Vincent's Hospital Melbourne, Fitzroy, Australia
- Belgium (3):
  - University Hospital Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Centre de Reference des Maladies Neuromusculaires et de la SLA - AP-HM Hopital de La Timone, Marseille
  - CHU de Nantes, Nantes
  - CHU de Nice - Hopital Pasteur 2 - Centre de reference des Maladies Neuromusculaires, Nice
  - AP-HP Hopital Pitie-Salpetriere, Paris
- Klinikum der Ludwig-Maximilians-Universitaet Muenchen, Munich, Germany
- Israel (2):
  - Hadassah University Hospital, Jerusalem
  - Schneider Children's Hospital of Israel, Petah Tikva
- Italy (3):
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Optimal Clinical Trials, Auckland, New Zealand
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - University College London Hospital, London
  - St. George's University Hospitals NHS Foundation Trust, London
  - Newcastle Freeman Hospital, Newcastle
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.edgewisetx.com